CLINICAL TRIAL: NCT05186688
Title: Braining Study - Implementation of Physical Activity for Patients and Staff in Specialist Psychiatry, Feasibility on Pilot Unit and Effect Evaluation in Randomized Controlled Multi-center Study.
Brief Title: Braining - Physical Exercise in Psychiatry - Evaluation of Feasibility, and Health Among Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Stockholm (Other Government)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Braining feasibility
Record Dates: First submitted 2021-12-25; First posted 2022-01-11 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-11

CONDITIONS: Mental Disorder
Keywords: physical exercise; mental disorders
MeSH Terms: conditions — Mental Disorders; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physical activity (Experimental): Patients are encouraged to participate in physical exercise at the psychiatric unit
  Interventions: Behavioral: Braining

INTERVENTIONS:
Behavioral: Braining — "Braining" is a clinical invention that helps patients in psychiatry to start and execute physical exercise (PE) regularly in psychiatric care. The core components are basic moderate to vigorous aerobic group training session and motivational work led by the psychiatric staff. Braining is used as add-on treatment to regular psychiatric care and is included in the patient care plan.

SUMMARY:
Physical exercise (PE) shows beneficial effects on somatic and psychiatric symptoms. "Braining" is a clinical invention where psychiatric staff exercise together with patients to help patients start and execute PE regularly. In the present study the feasibility of the intervention will be evaluated, how Braining is perceived, and preliminary effects on health and physical activity among patients. The investigators hypothesize that patients' health and physical activity will increase after participation in Braining at the unit. Braining will be implemented at two psychiatric pilot units in Region Stockholm, Sweden. During 6 months patients will be included and treated in 12 weeks PE intervention periods. To measure feasibility patients will answer self-rating questionnaires and be invited to semi structured interviews after receiving the intervention. Health will be measured by physical examination and blood test as well as self-ratings of depression, anxiety, sleep, hypomania, and quality of life before the intervention, every 4 weeks during the intervention, post the intervention, and at follow-up 12 months post the intervention. Physical activity will be rated before, during, after the intervention and at follow-up 12 months post the intervention using International Physical Activity Questionnaires (IPAQ) and Actigraph. All patients that fulfill inclusion criteria at the units will be invited to participate in the study, approximately 50 individuals in total.

DETAILED DESCRIPTION:
"Braining" is a clinical invention that helps patients in psychiatry to start and execute physical exercise (PE) regularly in psychiatric care. The core components are basic moderate to vigorous aerobic group training sessions and motivational work led by the psychiatric staff. Braining is used as add-on treatment to regular psychiatric care and is included in the patient care plan. Braining is unique in that it:

1. Includes trained psychiatric clinical staff exercising together with patients from both out- and inpatient ward units in daily, moderate to vigorous aerobic group training sessions
2. is included in regular healthcare fee, (free of charge)
3. includes a motivational and educational visit (as a group seminar or as an individual visit) at the start and end of a twelve-week exercise intervention
4. includes regular measurements (self-assessment questionnaires, blood samples, physical and mental health examination and education before and after the twelve-week exercise intervention)
5. offers short individual motivating visits before every training session, including assessment of day shape and fitness to participate.

In the present study focus is on the feasibility of the intervention, how Braining is perceived, and preliminary effects on health and physical activity among patients. The research questions are:

1. How do patients experience Braining in regards such as feasibility, acceptability, credibility, and effects on health and quality of life?
2. How do patients comply to Braining regarding completed training sessions and measurements?
3. What preliminary effect does Braining have on mental and physical health, quality of life and level of function in participating patients before compared to after short- and long-term exposure?

Examined from the following points of view:

* psychiatric symptoms, such as depression, hypomania, anxiety, insomnia?
* Somatic symptoms, such as blood pressure, resting heart rate, BMI, waist circumference, occurrence of somatic co-morbidity? Braining is to be implemented at 2 psychiatric care units starting nov 2021. Approximately 50 patients will be included. Planned design is an open trial study with monthly measurements during ongoing intervention (weeks 1, 4, 8 and 12) and one follow-up (12 months post inclusion). Physical activity level is measured with Actigraph and IPAQ 1 week before, 6 weeks in, after the intervention and at follow up.

Patients´ experience of Braining is examined with self-assessments and in interviews after the end of the intervention. Data analysis Qualitative analysis: Recorded material from interviews is transcribed and analyzed based on the thematic analysis method according to Braun & Clarke et al 2006). The method aims to understand the individual's perspective in relation to a particular phenomenon and is often used as an inductive hypothesis-generating approach. Continuous data will be analyzed using mixed effects models or t-test, nominal data analyzed mainly with chi2 test. In mixed effects models of differences between groups the interaction effect of group and time will be the central estimate.

ELIGIBILITY:
Inclusion Criteria:

* Patient at the psychiatric unit

Exclusion Criteria:

* Severe mental disorder such as ongoing mania, psychosis, and conditions when high risk of suicide or high risk of violence available according to the assessment of psychiatric staff at the unit.
* Medical conditions such as heart or lung disease, infection, abstinence where heart rate-increasing physical activity is considered contraindicated due to Medical reasons.
* Physical disability that makes it impossible to move independently to the gym and performing the indicated exercise in the training sessions.
* Mental disability which means that you can not participate in group training.
* Difficulty speaking or understanding the Swedish language.
* Ongoing heavy substance use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-03-02 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Actigraph GT3x | Change from inclusion to follow up 3 months after inclusion
  Objectively measured physical activity and sedentary time: Total physical activity as counts/day and time spent in sedentary, low, moderate and vigorous intensity as min/day.
Actigraph GT3x | At follow up 12 months after intervention.
  Objectively measured physical activity and sedentary time: Total physical activity as counts/day and time spent in sedentary, low, moderate and vigorous intensity as min/day.
International Physical Activity Questionnaires (IPAQ) | Change from inclusion to follow up 3 months after inclusion
  Self-reported physical activity: Total physical activity as Metabolic Energy Turnover (MET)hours/week and three level categories (low, moderate and high).
International Physical Activity Questionnaires (IPAQ) | At follow up 12 months after intervention.
  Self-reported physical activity: Total physical activity as Metabolic Energy Turnover (MET)hours/week and three level categories (low, moderate and high).
Patient Health Questionnaire 9 (PHQ-9) | Change from inclusion to follow up 3 months after inclusion
  Self rated depressive symptoms. Minimum value 0, maximum value 27, where higher values indicate more depressive symptoms.
Patient Health Questionnaire 9 (PHQ-9) | At follow up 12 months after intervention.
  Self rated depressive symptoms. Minimum value 0, maximum value 27, where higher values indicate more depressive symptoms.
Alcohol Use Disorders Identification Test AUDIT | Change from inclusion to follow up 3 months after inclusion
  Self rated alcohol use. Minimum value 0, maximum value 32, where higher values indicate higher alcohol use.
Alcohol Use Disorders Identification Test AUDIT | At follow up 12 months after intervention.
  Self rated alcohol use. Minimum value 0, maximum value 32, where higher values indicate higher alcohol use.
Drug Use Disorders Identification Test DUDIT | Change from inclusion to follow up 3 months after inclusion
  Self rated drug use. Minimum value 0, maximum value 44, where higher values indicate higher drug use.
Drug Use Disorders Identification Test DUDIT | At follow up 12 months after intervention.
  Self rated drug use. Minimum value 0, maximum value 44, where higher values indicate higher drug use.
Brunnsviken Brief Quality of Life Questionnaire (BBQ) | Change from inclusion to follow up 3 months after inclusion
  Self rated quality of life. Minimum value 0, maximum value 96, where higher values indicate higher quality of life satisfaction.
Brunnsviken Brief Quality of Life Questionnaire (BBQ) | At follow up 12 months after intervention.
  Self rated quality of life. Minimum value 0, maximum value 96, where higher values indicate higher quality of life satisfaction.
Acceptability of treatment among patients | At follow up 3-5 months after inclusion
  Semi-structured interviews
The Credibility/Expectancy Questionnaire (CEQ) | Week 1 of treatment
  Self rated Credibility of treatment. Minimum value 3, maximum value 27 for each factor, where higher values indicate greater Credibility/Expectancy of the treatment.
The Client Satisfaction Questionnaire-8 (CSQ-8) | post treatment, 12 weeks after enrollment
  Self rated satisfaction of treatment. Minimum value 8, maximum value 32 where higher values indicate greater satisfaction with the treatment.

SECONDARY OUTCOMES:
Generalised Anxiety Disorder 7-item scale (GAD-7) | Change from inclusion to follow up 3 months after inclusion
  Self rated anxiety symptoms. Minimum value 0, maximum value 21, where higher values indicate more anxiety symptoms.
Generalised Anxiety Disorder 7-item scale (GAD-7) | At follow up 12 months after intervention.
  Self rated anxiety symptoms. Minimum value 0, maximum value 21, where higher values indicate more anxiety symptoms.
Insomnia Severity Index (ISI) | Change from inclusion to follow up 3 months after inclusion
  Self rated insomnia symptoms. Minimum value 0, maximum value 28, where higher values indicate more insomnia symptoms.
Insomnia Severity Index (ISI) | At follow up 12 months after intervention.
  Self rated insomnia symptoms. Minimum value 0, maximum value 28, where higher values indicate more insomnia symptoms.
World health organization disability assessment schedule (WHODAS 2.0) | Change from inclusion to follow up 3 months after inclusion
  Self rated disability. Minimum value 0, maximum value 100, where higher values indicate more disability.
World health organization disability assessment schedule (WHODAS 2.0) | At follow up 12 months after intervention.
  Self rated disability. Minimum value 0, maximum value 100, where higher values indicate more disability.
Negative effects questionnaire (NEQ 20) | post treatment, 12 weeks after enrollment
  Self rated negative effects of treatment. Minimum value 0, maximum value 80, where higher values indicate more negative effects.
EuroQol (EQ-5D-5L) VAS | Change from inclusion to follow up 3 months after inclusion
  Self-assessment instrument for describing and valuing health. Defines health in terms of five dimensions: Mobility, Self-Care, Usual Activities, Pain/Discomfort, and Anxiety/Depression. Also included is an overall health rating on a 0-100 hash-marked, vertical visual analogue scale (EQ-VAS). Assessment the scores from the descriptive component can be reported as a five digit number ranging from 11111 (full health) to 55555 (worst health). A number of methods exist for analysing these five digit profiles. However, frequently they are converted to a single utility index using country specific value sets. A higher index number indicates a poorer self-assessed health.
EuroQol (EQ-5D-5L) VAS | At follow up 12 months after intervention.
  Self-assessment instrument for describing and valuing health. Defines health in terms of five dimensions: Mobility, Self-Care, Usual Activities, Pain/Discomfort, and Anxiety/Depression. Also included is an overall health rating on a 0-100 hash-marked, vertical visual analogue scale (EQ-VAS). Assessment the scores from the descriptive component can be reported as a five digit number ranging from 11111 (full health) to 55555 (worst health). A number of methods exist for analysing these five digit profiles. However, frequently they are converted to a single utility index using country specific value sets. A higher index number indicates a poorer self-assessed health.
Affective Self Rating Scale (AS-18) | Change from inclusion to follow up 3 months after inclusion
  Self-assessment of symptoms of depression and hypomania/mania. 9 items for depression and 9 items for mania. Score 0-72. A score of over 10 on the depressive or manic/hypomanic subscale should give rise to suspicion of ongoing depression and hypomania/mania respectively. Scores of over 10 on both the depressive and manic/hypomanic scale at the same time give may indicate an affective mixed state.
Affective Self Rating Scale (AS-18) | At follow up 12 months after intervention.
  Self-assessment of symptoms of depression and hypomania/mania. 9 items for depression and 9 items for mania. Score 0-72. A score of over 10 on the depressive or manic/hypomanic subscale should give rise to suspicion of ongoing depression and hypomania/mania respectively. Scores of over 10 on both the depressive and manic/hypomanic scale at the same time give may indicate an affective mixed state.
Blood pressure | Change from inclusion to follow up 3 months after inclusion
  systolic and diastolic, mmHg
Blood pressure | At follow up 12 months after intervention.
  systolic and diastolic, mmHg
Body mass index (BMI) | Change from inclusion to follow up 3 months after inclusion
  Weight in kg divided by the square of height in m
Body mass index (BMI) | At follow up 12 months after intervention.
  Weight in kg divided by the square of height in m
Waist circumference | Change from inclusion to follow up 3 months after inclusion
  Waist circumference, cm
Waist circumference | At follow up 12 months after intervention.
  Waist circumference, cm
Heart rate (HR) | Change from inclusion to follow up 3 months after inclusion
  Heart rate, beats per minute
Heart rate (HR) | At follow up 12 months after intervention.
  Heart rate, beats per minute
fasting blood sugar (FBS) | Change from inclusion to follow up 3 months after inclusion
  fasting blood sugar, mmol/l
fasting blood sugar (FBS) | At follow up 12 months after intervention.
  fasting blood sugar, mmol/l
Hemoglobin A1c (HbA1c) | Change from inclusion to follow up 3 months after inclusion
  Glycated hemoglobin, mmol/mol
hemoglobin A1c (HbA1c) | At follow up 12 months after intervention.
  Glycated hemoglobin, mmol/mol
Blood lipids | Change from inclusion to follow up 3 months after inclusion
  Total cholesterol, LDL cholesterol, HDL cholesterol, triglycerides, mmol/L
Blood lipids | At follow up 12 months after intervention.
  Total cholesterol, LDL cholesterol, HDL cholesterol, triglycerides, mmol/L
C-reactive protein (CRP) | Change from inclusion to follow up 3 months after inclusion
  Measurement of inflammation and infection, mmol/L
C-reactive protein (CRP) | At follow up 12 months after intervention.
  Measurement of inflammation and infection, mmol/L
Treatment Inventory of costs in patients with psychiatric disorders (TIC-P) | Change from inclusion to follow up 3 months after inclusion
  Work and illness measured by section C of Treatment Inventory of Costs in Patients with psychiatric disorders (TIC-P)
Treatment Inventory of costs in patients with psychiatric disorders (TIC-P) | At follow up 12 months after intervention.
  Work and illness measured by section C of Treatment Inventory of Costs in Patients with psychiatric disorders (TIC-P)
Thyroid releasing hormone (TSH) | Change from inclusion to follow up 3 months after inclusion
  Measurement of thyroid function, mUnits/L
Thyroid releasing hormone (TSH) | At follow up 12 months after intervention.
  Thyroid releasing hormone, measurement of thyroid function, mUnits/L
Complete blood count | Change from inclusion to follow up 3 months after inclusion
  The number of leukocytes, platelets and erythrocytes per unit volume in a sample of venous blood. Includes measurement of the hemoglobin, hematocrit and erythrocyte indices.
Complete blood count | At follow up 12 months after intervention.
  The number of leukocytes, platelets and erythrocytes per unit volume in a sample of venous blood. Includes measurement of the hemoglobin, hematocrit and erythrocyte indices.
Blood liver function test | Change from inclusion to follow up 3 months after inclusion
  Alanine transaminase (ALT) µkat/L, aspartate transaminase (AST) µkat/L, alkaline phosphatase (ALP) µkat/L albumin g/L, bilirubin µmol/L, gamma-glutamyltransferase (GGT) µkat/L, L-lactate dehydrogenase (LD) µkat/L
Blood liver function test | At follow up 12 months after intervention.
  Alanine transaminase (ALT) µkat/L, aspartate transaminase (AST) µkat/L, alkaline phosphatase (ALP) µkat/L albumin g/L, bilirubin µmol/L, gamma-glutamyltransferase (GGT) µkat/L, L-lactate dehydrogenase (LD) µkat/L

CONTACTS AND LOCATIONS:
Locations (1):
- Region Stockholm, Liljeholmsberget, Stockholm, Sweden